CLINICAL TRIAL: NCT01695239
Title: A Multicenter, Randomized, Double-Blind, Active and Placebo-Controlled 24-Week Study Followed by Long Term Evaluation of Efficacy and Safety of Ixekizumab (LY2439821) in Biologic Disease-Modifying Antirheumatic Drug-Naive Patients With Active Psoriatic Arthritis
Brief Title: A Study of Ixekizumab in Participants With Active Psoriatic Arthritis
Acronym: SPIRIT-P1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13731; I1F-MC-RHAP (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Results first posted 2016-10-27 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Psoriasis, Arthritic
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — ixekizumab; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ixekizumab Q2W (Experimental): Administered by 80 milligram (mg) subcutaneous (SC) injection every 2 weeks (Q2W).
  Interventions: Drug: Ixekizumab
- Ixekizumab Q4W (Experimental): Administered by 80 mg SC injection every 4 weeks (Q4W).
  Interventions: Drug: Ixekizumab
- Placebo (Placebo Comparator): Placebo for ixekizumab and placebo for adalimumab administered by SC injection.
  Interventions: Drug: Placebo
- Adalimumab Q2W (Active Comparator): Administered by 40 mg SC injection Q2W.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Ixekizumab — Administered SC
  Other Names: LY2439821
  Arms: Ixekizumab Q2W; Ixekizumab Q4W
Drug: Placebo — Administered SC
  Arms: Placebo
Drug: Adalimumab — Administered SC
  Arms: Adalimumab Q2W

SUMMARY:
This study will assess the safety and efficacy of ixekizumab (LY2439821) compared to placebo in participants with active psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Presents with established diagnosis of active psoriatic arthritis for at least 6 months, and currently meets Classification for Psoriatic Arthritis (CASPAR) criteria
* Active psoriatic arthritis (PsA) defined as the presence of at least 3 tender and at least 3 swollen joints
* Presence of active psoriatic skin lesion or a personal history of plaque psoriasis (Ps)
* Men must agree to use a reliable method of birth control or remain abstinent during the study
* Women must agree to use reliable birth control or remain abstinent during the study and for at least 12 weeks after stopping treatment

Exclusion Criteria:

* Current or prior use of biologic agents for treatment of Ps or PsA
* Inadequate response to greater than or equal to 4 conventional disease-modifying antirheumatic drugs (DMARDs)
* Current use of more than one conventional DMARD
* Evidence of active inflammatory arthritic syndromes or spondyloarthropathies other than PsA
* Have participated in any study with interleukin 17 (IL-17) antagonists, including ixekizumab
* Serious disorder or illness other than psoriatic arthritis
* Serious infection within the last 3 months
* Breastfeeding or nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (116):
- United States (37):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntsville, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tuscaloosa, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Upland, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trumbull, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boca Raton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orange Park, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zephyrhills, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Decatur, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marietta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cedar Rapids, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cumberland, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hagerstown, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Voorhees Township, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooklyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greensboro, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dayton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Duncansville, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orangeburg, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jackson, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kennewick, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clarksburg, West Virginia
- Belgium (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
- Bulgaria (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pleven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plovdiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sliven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sofia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stara Zagora
- Canada (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waterloo, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Québec
- Czechia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bruntál
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hlučín
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ostrava - Trebovice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zlín
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tallinn, Estonia
- France (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bordeaux
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nantes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orléans
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- Japan (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- Mexico (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis Potosí City
- Netherlands (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Almelo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maastricht
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nijmegen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sneek
- Poland (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Katowice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Środa Wielkopolska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- Russia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barnaul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kazan'
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petrozavodsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yekaterinburg
- Spain (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bilbao
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Majadahonda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sabadell
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santander
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
- Ukraine (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dnipropetrovsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Donetsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ivano-Frankivsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kharkiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lutsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lviv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Odesa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vinnytsia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zaporizhzhia
- United Kingdom (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cambridge, Cambridgeshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goodmayes, Essex
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Greater London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Headington, Oxford
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wolverhampton, West Midlands
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bradford, West Yorkshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds, West Yorkshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liverpool

REFERENCES:
- [Derived] Kristensen LE, McGonagle D, Rudwaleit M, Kameda H, Wurtzen PA, Ngantcha M, Holzkamper T, Smolen J. Synergistic Improvements in Synovitis, Enthesitis, and Patient-Reported Outcomes for Patients with Psoriatic Arthritis Treated with Ixekizumab in SPIRIT Trials. Rheumatol Ther. 2025 Apr;12(2):381-395. doi: 10.1007/s40744-025-00748-8. Epub 2025 Feb 27. PMID 40014255
- [Derived] Tillett W, Birt J, Vadhariya A, Ross S, Ngantcha M, Ng KJ. Filling the "GAP" in Real-World Assessment of Psoriatic Arthritis Disease Activity: Performance Characteristics of a Global/Pain Composite Endpoint. Rheumatol Ther. 2024 Oct;11(5):1101-1114. doi: 10.1007/s40744-024-00690-1. Epub 2024 Jul 2. PMID 38955921
- [Derived] Armstrong AW, Jaleel T, Merola JF, Gottlieb AB, Khattri S, Helt CC, Malatestinic WN, Ross SE, Ngantcha ME, de Vlam K. Ixekizumab Demonstrates Rapid and Consistent Efficacy for Patients with Psoriatic Arthritis, Regardless of Psoriasis Severity. Dermatol Ther (Heidelb). 2024 Jun;14(6):1615-1631. doi: 10.1007/s13555-024-01188-y. Epub 2024 May 30. PMID 38814433
- [Derived] Kameda H, Hagimori K, Morisaki Y, Holzkamper T, Konomi A, Dobashi H. Ixekizumab Efficacy in Patients with Severe Peripheral Psoriatic Arthritis: A Post Hoc Analysis of a Phase 3, Randomized, Double-Blind, Placebo-Controlled Study (SPIRIT-P1). Rheumatol Ther. 2023 Dec;10(6):1683-1703. doi: 10.1007/s40744-023-00605-6. Epub 2023 Oct 19. PMID 37858007
- [Derived] Coates LC, Smolen JS, Mease PJ, Husni ME, Merola JF, Lespessailles E, Kishimoto M, Macpherson L, Bradley AJ, Bolce R, Helliwell PS. Comparative performance of composite measures from two phase III clinical trials of ixekizumab in psoriatic arthritis. RMD Open. 2022 Sep;8(2):e002457. doi: 10.1136/rmdopen-2022-002457. PMID 36171019
- [Derived] Eder L, Tony HP, Odhav S, Agirregoikoa EG, Korkosz M, Schwartzman S, Sprabery AT, Gellett AM, Park SY, Bertram CC, Ogdie A. Responses to Ixekizumab in Male and Female Patients with Psoriatic Arthritis: Results from Two Randomized, Phase 3 Clinical Trials. Rheumatol Ther. 2022 Jun;9(3):919-933. doi: 10.1007/s40744-022-00445-w. Epub 2022 Apr 9. PMID 35397092
- [Derived] Deodhar AA, Combe B, Accioly AP, Bolce R, Zhu D, Gellett AM, Sprabery AT, Burmester GR. Safety of ixekizumab in patients with psoriatic arthritis: data from four clinical trials with over 2000 patient-years of exposure. Ann Rheum Dis. 2022 Jul;81(7):944-950. doi: 10.1136/annrheumdis-2021-222027. Epub 2022 Apr 7. PMID 35393269
- [Derived] Combe B, Tsai TF, Huffstutter JE, Sprabery AT, Lin CY, Park SY, Kronbergs A, Hufford MM, Nash P. Ixekizumab, with or without concomitant methotrexate, improves signs and symptoms of PsA: week 52 results from Spirit-P1 and Spirit-P2 studies. Arthritis Res Ther. 2021 Jan 27;23(1):41. doi: 10.1186/s13075-020-02388-5. PMID 33499913
- [Derived] Schweikert B, Malmberg C, Nunez M, Dilla T, Sapin C, Hartz S. Cost-effectiveness analysis of ixekizumab versus secukinumab in patients with psoriatic arthritis and concomitant moderate-to-severe psoriasis in Spain. BMJ Open. 2020 Aug 13;10(8):e032552. doi: 10.1136/bmjopen-2019-032552. PMID 32792421
- [Derived] Chandran V, van der Heijde D, Fleischmann RM, Lespessailles E, Helliwell PS, Kameda H, Burgos-Vargas R, Erickson JS, Rathmann SS, Sprabery AT, Birt JA, Shuler CL, Gallo G. Ixekizumab treatment of biologic-naive patients with active psoriatic arthritis: 3-year results from a phase III clinical trial (SPIRIT-P1). Rheumatology (Oxford). 2020 Oct 1;59(10):2774-2784. doi: 10.1093/rheumatology/kez684. PMID 32031665
- [Derived] Combe B, Rahman P, Kameda H, Canete JD, Gallo G, Agada N, Xu W, Genovese MC. Safety results of ixekizumab with 1822.2 patient-years of exposure: an integrated analysis of 3 clinical trials in adult patients with psoriatic arthritis. Arthritis Res Ther. 2020 Jan 21;22(1):14. doi: 10.1186/s13075-020-2099-0. PMID 31964419
- [Derived] Tillett W, Lin CY, Zbrozek A, Sprabery AT, Birt J. A Threshold of Meaning for Work Disability Improvement in Psoriatic Arthritis Measured by the Work Productivity and Activity Impairment Questionnaire. Rheumatol Ther. 2019 Sep;6(3):379-391. doi: 10.1007/s40744-019-0155-5. Epub 2019 Jun 1. PMID 31154634
- [Derived] Coates LC, Orbai AM, Morita A, Benichou O, Kerr L, Adams DH, Shuler CL, Birt J, Helliwell PS. Achieving minimal disease activity in psoriatic arthritis predicts meaningful improvements in patients' health-related quality of life and productivity. BMC Rheumatol. 2018 Aug 13;2:24. doi: 10.1186/s41927-018-0030-y. eCollection 2018. PMID 30886974
- [Derived] Gladman DD, Orbai AM, Klitz U, Wei JC, Gallo G, Birt J, Rathmann S, Shrom D, Marzo-Ortega H. Ixekizumab and complete resolution of enthesitis and dactylitis: integrated analysis of two phase 3 randomized trials in psoriatic arthritis. Arthritis Res Ther. 2019 Jan 29;21(1):38. doi: 10.1186/s13075-019-1831-0. PMID 30696483
- [Derived] Gottlieb AB, Strand V, Kishimoto M, Mease P, Thaci D, Birt J, Lee CH, Shuler CL, Lin CY, Gladman DD. Ixekizumab improves patient-reported outcomes up to 52 weeks in bDMARD-naive patients with active psoriatic arthritis (SPIRIT-P1). Rheumatology (Oxford). 2018 Oct 1;57(10):1777-1788. doi: 10.1093/rheumatology/key161. PMID 29945203
- [Derived] Coates LC, Kishimoto M, Gottlieb A, Shuler CL, Lin CY, Lee CH, Mease PJ. Ixekizumab efficacy and safety with and without concomitant conventional disease-modifying antirheumatic drugs (cDMARDs) in biologic DMARD (bDMARD)-naive patients with active psoriatic arthritis (PsA): results from SPIRIT-P1. RMD Open. 2017 Dec 22;3(2):e000567. doi: 10.1136/rmdopen-2017-000567. eCollection 2017. PMID 29299340
- [Derived] van der Heijde D, Gladman DD, Kishimoto M, Okada M, Rathmann SS, Moriarty SR, Shuler CL, Carlier H, Benichou O, Mease PJ. Efficacy and Safety of Ixekizumab in Patients with Active Psoriatic Arthritis: 52-week Results from a Phase III Study (SPIRIT-P1). J Rheumatol. 2018 Mar;45(3):367-377. doi: 10.3899/jrheum.170429. Epub 2017 Dec 15. PMID 29247148
- [Derived] Mease PJ, van der Heijde D, Ritchlin CT, Okada M, Cuchacovich RS, Shuler CL, Lin CY, Braun DK, Lee CH, Gladman DD; SPIRIT-P1 Study Group. Ixekizumab, an interleukin-17A specific monoclonal antibody, for the treatment of biologic-naive patients with active psoriatic arthritis: results from the 24-week randomised, double-blind, placebo-controlled and active (adalimumab)-controlled period of the phase III trial SPIRIT-P1. Ann Rheum Dis. 2017 Jan;76(1):79-87. doi: 10.1136/annrheumdis-2016-209709. Epub 2016 Aug 23. PMID 27553214

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Double-Blind Treatment Period was Week 0 up to Week 24 (Inadequate responders (IR) Week 16-24) followed by the combined extension period and long-term extension period from Week 24 to Week 156.
Groups:
- Placebo (PBO): Participants received placebo for ixekizumab (ixe) as 2 subcutaneous (SC) injections and placebo for adalimumab as one SC injection for a total of 3 injections at Week 0. Placebo for ixekizumab and placebo for adalimumab were given as single SC injections every 2 weeks (Q2W) from Week 2 to Week 24.
- Adalimumab (ADA) Q2W: Participants received 40 mg of adalimumab as one SC injection and placebo for ixekizumab as 2 SC injections for a total of 3 injections at Week 0. Participants received one SC injection of 40 mg of adalimumab and one SC injection of placebo for ixekizumab Q2W from Week 2 to Week 24.
- Ixe Q4W: Participants received a starting dose of 160 mg of ixekizumab given as 2 SC injections of 80 mg and placebo for adalimumab as one SC injection for a total of 3 injections at Week 0. Participants received one SC injection of 80 mg of ixekizumab or placebo for ixekizumab Q2W from Week 2 to Week 24. Participants received one SC injection of placebo for adalimumab Q2W from Week 2 to Week 24.
- Ixe Q2W: Participants received a starting dose of 160 mg of ixekizumab given as 2 SC injections of 80 mg and placebo for adalimumab as one SC injection for a total of 3 injections at Week 0. Participants received one SC injection of 80 mg of ixekizumab Q2W from Week 2 to Week 24. Participants received one SC injection of placebo for adalimumab Q2W from Week 2 to Week 24.
- Inadequate Responders (IR)/Ixe Q4W: Placebo Week 16 inadequate responders (IRs) re-randomized to ixekizumab 80 mg every 4 weeks (Q4W) received a starting dose of 160 mg of ixekizumab given as 2 SC injections of 80 mg and placebo for adalimumab as one SC injection for a total of 3 injections at Week 16. Participants received one SC injection of 80 mg of ixekizumab or placebo for ixekizumab Q2W from Week 18 to Week 24. Participants received one SC injection of placebo for adalimumab Q2W from Week 18 to Week 24. Participants also received rescue therapy. Ixekizumab Q4W IRs received one SC injection of 80 mg of ixekizumab or placebo for ixekizumab Q2W from Week 18 to Week 24. Participants received one SC injection of placebo for adalimumab Q2W from Week 18 to Week 24. Participants also received rescue therapy.
- IR/Ixe Q2W: Placebo IRs re-randomized to ixekizumab 80 mg Q2W received a starting dose of 160 mg of ixekizumab given as 2 SC injections of 80 mg and placebo for adalimumab as one SC injection for a total of 3 injections at Week 16. Participants received one SC injection of 80 mg of ixekizumab Q2W from Week 18 to Week 24. Participants received one SC injection of placebo for adalimumab Q2W from Week 18 to Week 24. Participants also received rescue therapy. Ixekizumab 80 mg Q2W IRs received one SC injection of 80 mg of ixekizumab Q2W from Week 18 to Week 24. Participants received one SC injection of placebo for adalimumab Q2W from Week 18 to Week 24. Participants also received rescue therapy.
- IR PBO Washout: Adalimumab Q2W IRs re-randomized to ixekizumab 80 mg Q4W or ixekizumab 80 mg Q2W. Participants received 40 mg of adalimumab as one SC injection and placebo for ixekizumab as 2 SC injections for a total of 3 injections at Week 16. Placebo for ixekizumab and placebo for adalimumab were given as single SC injections Q2W from Week 18 to Week 22. Participants received a starting dose of 160 mg of ixekizumab given as 2 SC injections of 80 mg and placebo for adalimumab as one SC injection for a total of 3 injections at Week 24.
- PBO Washout: Adalimumab Q2W participants re-randomized to ixekizumab 80 mg Q4W or ixekizumab Q2W Week 24. Participants received 40 mg of adalimumab as one SC injection and placebo for ixekizumab as 2 SC injections for a total of 3 injections at Week 24. Placebo for ixekizumab and placebo for adalimumab were given as single SC injections Q2W from Week 26 to Week 30. Participants received a dose of 80 mg of ixekizumab given as 1 SC injection at Week 32.
- Ixe Q4W/Ixe Q4W: Participants continuing on 1 injection of ixekizumab 80 mg Q4W starting on Week 24 and ending on Week 156 alternating with placebo injections Q4W starting on Week 26 and ending on Week 154. Additionally, includes placebo washout participants who were re-randomized to ixekizumab 80 mg given at Week 24 followed by 1 SC injection of 80 mg of ixekizumab Q4W starting on Week 28 and ending on Week 156 alternating with placebo injections Q4W starting on Week 26 and ending on Week 154. Placebo washout participants who re-randomized at Week 24 receive 1 SC injection of 80 mg of ixekizumab Q4W starting on Week 32 and ending on Week 156 alternating with placebo injections Q4W starting on Week 34 and ending on Week 154.
- Ixe Q2W/Ixe Q2W: Participants continuing on 1 injection of ixekizumab 80 mg Q2W starting on Week 24 and ending on Week 156. Additionally, includes placebo washout participants who were re-randomized to ixekizumab 80 mg Q2W at Week 16 and Week 24. Placebo washout participants who re-randomized at Week 16 receive a starting dose of 160 mg ixekizumab given as 2 SC injections of 80 mg given at Week 24 followed by 1 SC injection of 80 mg of ixekizumab Q2W starting on Week 28 and ending on Week 156. Placebo washout participants who re-randomized at Week 24 receive 1 SC injection of 80 mg of ixekizumab Q2W starting on Week 32 and ending on Week 156.
- Placebo Post-Treatment Follow-up Period: Participants discontinued the study early and entered the post-treatment follow-up period. Participants received placebo immediately prior to entering the post-treatment follow-up period.
- Adalimumab Post-Treatment Follow-up Period: Participants discontinued the study early and entered the post-treatment follow-up period. Participants received adalimumab Q2W immediately prior to entering the post-treatment follow-up period.
- Ixekizumab 80mg Q4W Post-Treatment Follow-up Period: Participants either completed the study or discontinued the study early and entered the post-treatment follow-up period. Participants received ixekizumab 80 mg Q4W immediately prior to entering the post-treatment follow-up period.
- Ixekizumab 80mg Q2W Post-Treatment Follow-up Period: Participants either completed the study or discontinued the study early and entered the post-treatment follow-up period. Participants received ixekizumab 80 mg Q2W immediately prior to entering the post-treatment follow-up period.
Period: Double-Blind (DB) Treatment Period
Arm/Group | Placebo (PBO) | Adalimumab (ADA) Q2W | Ixe Q4W | Ixe Q2W | Inadequate Responders (IR)/Ixe Q4W | IR/Ixe Q2W | IR PBO Washout | PBO Washout | Ixe Q4W/Ixe Q4W | Ixe Q2W/Ixe Q2W | Placebo Post-Treatment Follow-up Period | Adalimumab Post-Treatment Follow-up Period | Ixekizumab 80mg Q4W Post-Treatment Follow-up Period | Ixekizumab 80mg Q2W Post-Treatment Follow-up Period
Started | 106 | 101 | 107 | 103 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 106 | 101 | 107 | 102 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Classified as Inadequate Responder (IR) | 27 | 9 | 11 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 91 | 97 | 97 | 96 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 15 | 4 | 10 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Entry Criteria Not Met | 1 | 1 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 4 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: IR Participants (Week 16 Up To Week 24)
Arm/Group | Placebo (PBO) | Adalimumab (ADA) Q2W | Ixe Q4W | Ixe Q2W | Inadequate Responders (IR)/Ixe Q4W | IR/Ixe Q2W | IR PBO Washout | PBO Washout | Ixe Q4W/Ixe Q4W | Ixe Q2W/Ixe Q2W | Placebo Post-Treatment Follow-up Period | Adalimumab Post-Treatment Follow-up Period | Ixekizumab 80mg Q4W Post-Treatment Follow-up Period | Ixekizumab 80mg Q2W Post-Treatment Follow-up Period
Started | 0 (Only inadequate responders were included.) | 0 (Only inadequate responders were included.) | 0 (Only inadequate responders were included.) | 0 (Only inadequate responders were included.) | 24 (IR from placebo who re-randomized to ixeQ4W and IR from ixeQ4W.) | 24 (IR from placebo who re-randomized to ixeQ2W and IR from ixeQ2W.) | 9 (Adalimumab Q2W (IR) who re-randomized to IxeQ2W or IxeQ4W and PBO for ixe and adalimumab.) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 24 | 24 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Placebo Washout (Week 24 Up To Week 32)
Arm/Group | Placebo (PBO) | Adalimumab (ADA) Q2W | Ixe Q4W | Ixe Q2W | Inadequate Responders (IR)/Ixe Q4W | IR/Ixe Q2W | IR PBO Washout | PBO Washout | Ixe Q4W/Ixe Q4W | Ixe Q2W/Ixe Q2W | Placebo Post-Treatment Follow-up Period | Adalimumab Post-Treatment Follow-up Period | Ixekizumab 80mg Q4W Post-Treatment Follow-up Period | Ixekizumab 80mg Q2W Post-Treatment Follow-up Period
Started | 0 | 0 | 0 | 0 | 0 (Only included PBO washout participants.) | 0 (Only included PBO washout participants.) | 0 (Only included PBO washout participants.) | 88 (Adalimumab Q2W responders who re-randomized to IxeQ2W or IxeQ4W and PBO for ixe and adalimumab.) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 77 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Entry Criteria Not Met | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Extension Long-Term Extension Periods
Arm/Group | Placebo (PBO) | Adalimumab (ADA) Q2W | Ixe Q4W | Ixe Q2W | Inadequate Responders (IR)/Ixe Q4W | IR/Ixe Q2W | IR PBO Washout | PBO Washout | Ixe Q4W/Ixe Q4W | Ixe Q2W/Ixe Q2W | Placebo Post-Treatment Follow-up Period | Adalimumab Post-Treatment Follow-up Period | Ixekizumab 80mg Q4W Post-Treatment Follow-up Period | Ixekizumab 80mg Q2W Post-Treatment Follow-up Period
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (Only included combined extension participants.) | 187 (IxeQ4W who re-randomized to ixeQ4W.) | 183 (IxeQ2W who re-randomized to ixeQ2W.) | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 121 | 122 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 66 | 61 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 37 | 31 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 21 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 7 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Post-Treatment Follow-Up Period
Arm/Group | Placebo (PBO) | Adalimumab (ADA) Q2W | Ixe Q4W | Ixe Q2W | Inadequate Responders (IR)/Ixe Q4W | IR/Ixe Q2W | IR PBO Washout | PBO Washout | Ixe Q4W/Ixe Q4W | Ixe Q2W/Ixe Q2W | Placebo Post-Treatment Follow-up Period | Adalimumab Post-Treatment Follow-up Period | Ixekizumab 80mg Q4W Post-Treatment Follow-up Period | Ixekizumab 80mg Q2W Post-Treatment Follow-up Period
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (Only included post-treatment follow-up participants.) | 0 (Only included post-treatment follow-up participants.) | 20 (Participants who discontinued early and received PBO.) | 1 (Participants who discontinued early and received adalimumab.) | 165 (IxeQ4W participants who entered post-treatment follow-up.) | 171 (IxeQ2W participants who entered post-treatment follow-up.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 0 | 156 | 166
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 9 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Placebo: Participants received placebo for ixekizumab as 2 SC injections and placebo for adalimumab as one SC injection for a total of 3 injections at Week 0. Placebo for ixekizumab and placebo for adalimumab were given as single SC injections Q2W from Week 2 to Week 24.
- ADA Q2W: Participants received 40 mg of adalimumab as one SC injection and placebo for ixekizumab as 2 SC injections for a total of 3 injections at Week 0. Participants received one SC injection of 40 mg of adalimumab and one SC injection of placebo for ixekizumab Q2W from Week 2 to Week 24.
- Total: Total of all reporting groups
Arm/Group | Placebo | ADA Q2W | Ixe Q4W | Ixe Q2W | Total
Number analyzed (Participants) | 106 | 101 | 107 | 103 | 417
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.60 (12.32) | 48.58 (12.43) | 49.07 (10.07) | 49.79 (12.62) | 49.52 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 50 | 62 | 55 | 225
  Male | 48 | 51 | 45 | 48 | 192
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 2 | 2 | 9
  Asian | 5 | 3 | 2 | 5 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 99 | 95 | 102 | 96 | 392
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 5 | 4 | 20
  Not Hispanic or Latino | 92 | 83 | 94 | 87 | 356
  Unknown or Not Reported | 8 | 13 | 8 | 12 | 41
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 9 | 7 | 10 | 8 | 34
  United States | 22 | 21 | 20 | 20 | 83
  Japan | 4 | 2 | 2 | 4 | 12
  Ukraine | 9 | 7 | 9 | 10 | 35
  United Kingdom | 3 | 5 | 5 | 4 | 17
  Spain | 4 | 2 | 3 | 4 | 13
  Canada | 1 | 1 | 2 | 0 | 4
  Czechia | 22 | 25 | 23 | 22 | 92
  Netherlands | 1 | 0 | 1 | 0 | 2
  Belgium | 2 | 2 | 0 | 1 | 5
  Poland | 16 | 14 | 15 | 15 | 60
  Mexico | 3 | 4 | 3 | 2 | 12
  France | 1 | 0 | 1 | 1 | 3
  Bulgaria | 3 | 4 | 5 | 4 | 16
  Estonia | 6 | 7 | 8 | 8 | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20 (ACR20) Response at Week 24 (Efficacy of Ixekizumab in Participants With Active Psoriatic Arthritis. Measure: American College of Rheumatology 20 Index [ACR20])
Description: ACR20 response is defined as a ≥20% improvement from baseline for tender joint count (TJC) and swollen joint count (SJC) and in at least 3 of the following 5 criteria: Participant's assessment of Joint Pain visual analog scale (VAS), Participant's Global Assessment of Disease Activity VAS (PatGA), Physician's Global Assessment of the Disease Activity VAS (PGA), Participant's Assessment of Physical Function using the Health Assessment Questionnaire Disability Index (HAQ-DI), or Acute Phase Reactant as measured by high sensitivity C-reactive protein (hs-CRP).
Time Frame: Week 24
Population: All randomized participants. Nonresponder Imputation (NRI) is applied for inadequate responders at Week 16 and participants who had missing data at Week 24 for any reason including discontinuation.
Measure: Number; unit: percentage of participants
Groups:
- Adalimumab Q2W: Participants received 40 mg of adalimumab as one SC injection and placebo for ixekizumab as 2 SC injections for a total of 3 injections at Week 0. Participants received one SC injection of 40 mg of adalimumab and one SC injection of placebo for ixekizumab Q2W from Week 2 to Week 24.
- Ixekizumab Q4W: Participants received a starting dose of 160 mg of ixekizumab given as 2 SC injections of 80 mg and placebo for adalimumab as one SC injection for a total of 3 injections at Week 0. Participants received one SC injection of 80 mg of ixekizumab or placebo for ixekizumab Q2W from Week 2 to Week 24. Participants received one SC injection of placebo for adalimumab Q2W from Week 2 to Week 24.
- Ixekizumab Q2W: Participants received a starting dose of 160 mg of ixekizumab given as 2 SC injections of 80 mg and placebo for adalimumab as one SC injection for a total of 3 injections at Week 0. Participants received one SC injection of 80 mg of ixekizumab Q2W from Week 2 to Week 24. Participants received one SC injection of placebo for adalimumab Q2W from Week 2 to Week 24.
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 106 | 101 | 107 | 103
percentage of participants | 30.2 | 57.4 | 57.9 | 62.1
Statistical Analysis 1: Comparison: Placebo vs Adalimumab Q2W; Test type: Superiority or Other; p < 0.001, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab Q4W; Test type: Superiority or Other; p < 0.001, Regression, Logistic
Statistical Analysis 3: Comparison: Placebo vs Ixekizumab Q2W; Test type: Superiority or Other; p < 0.001, Regression, Logistic

2. Secondary Outcome: Percentage of Participants Achieving ACR20 Response
Description: ACR20 response is defined as a ≥20% improvement from baseline for TJC and SJC and in at least 3 of the following 5 criteria: Participant's assessment of Joint Pain VAS, Participant's Global Assessment of Disease Activity VAS, Physician's Global Assessment of the Disease Activity VAS, Participant's Assessment of Physical Function using the HAQ-DI, or hs-CRP.
Time Frame: Week 12
Population: All randomized participants. NRI is applied for inadequate responders at Week 16 and participants who had missing data at Week 24 for any reason including discontinuation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 106 | 101 | 107 | 103
percentage of participants | 31.1 | 51.5 | 57.0 | 60.2

3. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50 (ACR50) Response
Description: ACR50 response is defined as a ≥50% improvement from baseline for TJC and SJC and in at least 3 of the following 5 criteria: Participant's assessment of Joint Pain VAS, Participant's Global Assessment of Disease Activity VAS, Physician's Global Assessment of the Disease Activity VAS, Participant's Assessment of Physical Function using the HAQ-DI, or hs-CRP.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 106 | 101 | 107 | 103
percentage of participants | 15.1 | 38.6 | 40.2 | 46.6

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70 (ACR70) Score
Description: ACR70 response is defined as a ≥70% improvement from baseline for TJC and SJC and in at least 3 of the following 5 criteria: Participant's assessment of Joint Pain VAS, Participant's Global Assessment of Disease Activity VAS, Physician's Global Assessment of the Disease Activity VAS, Participant's Assessment of Physical Function using the HAQ-DI, or hs-CRP.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 106 | 101 | 107 | 103
percentage of participants | 5.7 | 25.7 | 23.4 | 34.0

5. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Scores (Quality of Life and Outcome Assessments Measures: Participant Reported Outcomes [PRO])
Description: HAQ-DI is a participant reported questionnaire that measures disease-associated disability (physical function). It consists of 24 questions with 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and other daily activities. The disability section scores the participant's self-perception on the degree of difficulty (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do), covering the 8 domains. The HAQ-DI is a composite ranging from 0-3 with lower scores indicating less functional disability. The reported use of special aids or devices and/or the need for assistance of another person to perform these activities is assessed. Least Square (LS) mean was calculated using Mixed Model Repeated Measurements (MMRM) analysis with treatment, baseline score, geographic region, baseline conventional disease modifying anti-rheumatic drugs (cDMARD) experience, visit, and treatment-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants with baseline and post baseline HAQ-DI data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 105 | 97 | 103 | 98
units on a scale | -0.1797 (0.0524) | -0.3712 (0.0510) | -0.4431 (0.0503) | -0.4963 (0.0507)

6. Secondary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS) (Efficacy of Ixekizumab in Participants With Active Psoriatic Arthritis. Measure: Modified Total Sharp Score [mTSS])
Description: The mTSS measures the extent of bone erosions (20 joints per hand and 12 joints per foot) and joint space narrowing (20 joints per hand and 6 joints per foot), with higher scores representing greater damage. An increase from baseline represents disease progression and / or joint worsening. Scores range from 0-528. LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, and baseline cDMARD experience, visit, treatment by visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants with baseline and post baseline mTSS data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 106 | 101 | 107 | 103
units on a scale | 0.49 (0.086) | 0.10 (0.085) | 0.17 (0.082) | 0.08 (0.083)

7. Secondary Outcome: Percentage of Participants Achieving Psoriasis Area and Severity Index 75%, 90%, 100% (PASI 75, 90, 100)
Description: The PASI is an index that combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of desquamation, erythema, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no psoriasis to 72 for the most severe disease. Participants achieving PASI 75 were defined as having an improvement of at least 75% in the PASI compared to their baseline measures. Participants achieving PASI 90 were defined as having an improvement of ≥90% in the PASI score compared to baseline. Participants achieving PASI 100 were defined as having an improvement of 100% in the PASI score compared to baseline.
Time Frame: Week 12
Population: All randomized participants with baseline psoriatic lesion(s) involving ≥3% BSA. NRI is applied for inadequate responders at Week 16 and participants who had missing data at Week 24 for any reason including discontinuation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 67 | 68 | 73 | 59
percentage of participants
  PASI 75 | 7.5 | 33.8 | 75.3 | 69.5
  PASI 90 | 1.5 | 22.1 | 52.1 | 57.6
  PASI 100 | 1.5 | 14.7 | 31.5 | 40.7

8. Secondary Outcome: Change From Baseline in Leeds Enthesitis Index (LEI)
Description: The LEI was developed specifically for use in PsA. It measures enthesitis at 6 sites (lateral epicondyle, left and right; medial femoral condyle, left and right; Achilles tendon insertion, left and right). Each site was assigned a score of 0 (absent) or 1 (present); the results from each site were then added to produce a total score (range 0 to 6). LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, baseline cDMARD experience, visit, treatment by visit interaction.
Time Frame: Baseline, Week 12
Population: All randomized participants who had baseline enthesitis, baseline LEI score and post baseline LEI score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 57 | 55 | 70 | 56
units on a scale | -0.8 (0.24) | -0.8 (0.24) | -0.9 (0.21) | -1.5 (0.24)

9. Secondary Outcome: Change From Baseline in Itching Severity Using the Itch Numeric Rating Scale (NRS) (Quality of Life and Outcome Assessments Measures: Participant Reported Outcomes [PRO])
Description: The Itch NRS is a participant-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participant's itching from psoriasis was indicated by circling the number that best described the worst level of itching in the past 24 hours. LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, baseline cDMARD experience, visit, and treatment-by-visit interaction.
Time Frame: Baseline, Week 12
Population: All randomized participants who had baseline psoriatic lesion(s) involving >=3% BSA, baseline itch NRS score and post baseline itch NRS score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 67 | 68 | 73 | 59
units on a scale | 0.2 (0.27) | -1.4 (0.28) | -2.6 (0.27) | -2.8 (0.30)

10. Secondary Outcome: Change From Baseline in Fatigue Severity NRS Score (Quality of Life and Outcome Assessments Measures: Participant Reported Outcomes [PRO])
Description: The Fatigue Severity NRS is a participant-administered single-item 11-point horizontal scale anchored at 0 and 10, with 0 representing "no fatigue" and 10 representing "as bad as you can imagine." Participants rated their fatigue (feeling tired or worn out) by circling the 1 number that described their worst level of fatigue during the past 24 hours. LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, baseline cDMARD experience, visit, and treatment-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants who had baseline and post baseline fatigue NRS data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 103 | 97 | 101 | 97
units on a scale | -1.3 (0.25) | -1.5 (0.24) | -1.6 (0.24) | -1.9 (0.24)

11. Secondary Outcome: Change From Baseline in Joint Space Narrowing Score (JSN) And Bone Erosion Score (BES)
Description: JSN score (a component of the modified Total Sharp Score [mTSS]) measures the extent of joint space narrowing in peripheral joints. JSN (20 joints per hand and 6 joints per foot), with higher scores representing greater damage. JSN score range is 0 (no narrowing) to 208 (high narrowing). Increase from baseline represents disease progression and / or joint worsening. BES (a component of the [mTSS]) measures the extent of bone erosion in peripheral joints. BES measures the extent of joint erosions (20 joints per hand and 12 joints per foot), with higher scores representing greater damage. Erosion score range is from 0 (no erosion) to 320 (high erosion). LS mean was calculated using linear extrapolation for ANCOVA analysis with treatment, baseline score, geographic region, and baseline cDMARD experience.
Time Frame: Baseline, Week 24
Population: All randomized participants who had baseline and post baseline JSN data. All randomized participants who had baseline and post baseline BES data. Linear extrapolation was used to impute missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 91 | 95 | 97 | 96
units on a scale
  Joint Space Narrowing Score | 0.07 (0.031) | 0.01 (0.031) | 0.04 (0.030) | 0.01 (0.030)
  Bone Erosion Score | 0.44 (0.077) | 0.12 (0.077) | 0.15 (0.075) | 0.08 (0.075)

12. Secondary Outcome: Change From Baseline in Medical Outcomes Study 36-item Short Form Health Survey (SF-36): Physical Component Summary (PCS) and Mental Component Summary (MCS) (Quality of Life and Outcome Assessments Measures: Participant Reported Outcomes [PRO])
Description: SF-36 is a standardized participant-administered measure designed to evaluate 8 domains of functional health and well being: physical and social functioning, physical and emotional role (role-physical, role-emotional) limitations, bodily pain, general health, vitality, mental health with 2 components (physical component score [PCS] and mental component score [MCS]). The PCS and MCS scores range from 0 to 100, with higher scores indicating better levels of function and/or better health. LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, baseline cDMARD experience, visit, and treatment-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants who had baseline and post baseline PCS data. All randomized participants who had baseline and post baseline MCS data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 99 | 95 | 98 | 95
units on a scale
  PCS Score | 2.94 (0.958) | 6.78 (0.904) | 7.45 (0.894) | 8.24 (0.898)
  MCS Score | 2.67 (1.013) | 4.22 (0.943) | 4.86 (0.933) | 3.39 (0.936)

13. Secondary Outcome: Change From Baseline in Quick Inventory of Depressive Symptomatology-Self Reported 16 Items (QIDS-SR16) (Quality of Life and Outcome Assessments. Measures: Patient Reported Outcomes [PRO])
Description: The QIDS-SR16 is a self-administered 16-item instrument intended to assess the existence and severity of symptoms of depression. A participant is asked to consider each statement as it relates to the way they have felt for the past 7 days. Each item scaled from 0 (no symptoms) to 3 (all symptoms). The 16 items corresponding to 9 depression domains are summed to give a single score ranging from 0 to 27, with higher scores denoting greater symptom severity. LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, baseline cDMARD experience, visit, and treatment-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants who had baseline and post baseline QIDS-SR16 data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 101 | 98 | 102 | 99
units on a scale | -0.9 (0.36) | -1.6 (0.33) | -0.8 (0.32) | -0.7 (0.32)

14. Secondary Outcome: Change From Baseline in Disease Activity Score (28 Diarthrodial Joint Count) Based on C-ReactiveProtein (DAS28-CRP) Measure: Non-Arthritic Disease
Description: The DAS28-CRP is a measure of disease activity in 28 joints that consists of a composite numerical score with the following variables: TJC28, SJC28, hs-CRP measured in milligram/liter (mg/L), and Participant's Global Assessment of Disease Activity recorded by participants on a 0 to 100 millimeter (mm) VAS. For DAS28-CRP, the Tender Joint Count 28 (TJC28) and Swollen Joint Count (SJC28) are a subset of TJC and SJC, and include 14 joints on each side of the body: 2 shoulders, 2 elbows, 2 wrists, 10 metacarpophalangeal joints, the 2 interphalangeal joints of the thumb, the 8 proximal interphalangeal joints, and the 2 knees. DAS28 values range from 0 to 9.4. Higher values indicate more severe symptoms and greater functional impairment. LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, baseline cDMARD experience, visit, and treatment-by-visit.
Time Frame: Baseline, Week 24
Population: All randomized participants who had baseline and post baseline DAS28-CRP data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 104 | 99 | 106 | 99
units on a scale | -0.835 (0.1307) | -1.743 (0.1215) | -1.955 (0.1206) | -2.036 (0.1225)

15. Secondary Outcome: Percentage of Participants Meeting the Psoriatic Arthritis Response Criteria (PsARC Modified)
Description: The PsARC is a composite criteria reported in terms of the percentage of participants achieving response according to the following criterion: TJC, SJC, PGA, and PatGA. Overall response is defined by improvement from baseline assessment in 2 of 4 criteria, 1 of which must be a joint count; there must not be worsening in any of the 4 criteria: at least 30% reduction in TJC, at least 30% reduction in SJC, at least a 20 millimeter (mm) reduction in PGA and at least a 20 mm reduction in PatGA which is equivalent to 20 mm reduction. The results from the 2 VAS measures were assessed as a difference from baseline in mm.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 106 | 101 | 107 | 103
percentage of participants | 32.1 | 58.4 | 57.9 | 66.0

16. Secondary Outcome: Percentage of Participants Achieving Static Physician Global Assessment (sPGA) of 0 or 1 and With at Least a 2-point Improvement From Baseline
Description: The sPGA is the physician's determination of the severity of the participant's psoriasis lesions overall at a given time point. Overall lesions were categorized by descriptions for induration, erythema, and scaling. For the analysis of responses, the participant's psoriasis was assessed at a given time point on in which 0 = clear, 1 = minimal, 2 = mild, 3 = moderate, 4 = severe, 5 = very severe.
Time Frame: Week 24
Population: All randomized participants who have plaque psoriasis and sPGA ≥3 at baseline. NRI is applied for inadequate responders at Week 16 and participants who had missing data at Week 24 for any reason including discontinuation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 41 | 37 | 52 | 41
percentage of participants | 17.1 | 62.2 | 65.4 | 73.2

17. Secondary Outcome: Percent Change From Baseline in Body Surface Area (BSA)
Description: The investigator evaluated the percentage involvement of psoriasis on each participant's BSA on a continuous scale from 0% = no involvement to 100% = full involvement, where 1% corresponded to the size of the participant's handprint including the palm, fingers, and thumb. LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, baseline cDMARD experience, visit, and treatment-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants who have plaque psoriasis at baseline and who had baseline and post baseline BSA data.
Measure: Least Squares Mean (Standard Error); unit: percent change in BSA
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 99 | 94 | 100 | 91
percent change in BSA | -2.7 (1.36) | -9.5 (1.35) | -12.0 (1.32) | -10.6 (1.39)

18. Secondary Outcome: Change From Baseline in the Nail Psoriasis Severity Index (NAPSI) Score Fingernail Involvement at Baseline
Description: The NAPSI scale is used to evaluate the severity of fingernail bed Ps and fingernail matrix Ps by area of involvement. The fingernail is divided into quadrants. Each fingernail is given a score for fingernail bed Ps 0 (none) to 4 (Ps in 4 quadrants of the fingernail) and fingernail matrix Ps 0 (none) to 4 (Ps in 4 quadrants of the matrix), depending on the presence (score of 1) or absence (score of 0) of any of the features of fingernail bed or matrix Ps in each quadrant. The sum of all fingernails equals the total NAPSI score range is from 0 (no effect) to 80 (more severe psoriasis). LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, baseline cDMARD experience, visit, and treatment-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants who had baseline fingernail involvement, baseline NAPSI score and post baseline NAPSI score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 69 | 68 | 66 | 69
units on a scale | -2.4 (1.66) | -10.7 (1.49) | -14.0 (1.54) | -15.5 (1.49)

19. Secondary Outcome: Change From Baseline in Leeds Dactylitis Index-Basic (LDI-B)
Description: The LDI-B measures the severity of dactylitis. In each digit, the ratio of the circumference of the affected digit to the circumference of the digit on the opposite hand or foot measured in mm. Each dactylitic digit was defined by a minimum increase of 10% in circumference over the contra-lateral digit. If the same digits on each hand or foot were thought to be involved, the clinician referred to a table of normative values for a value which was used to provide the comparison. The calculated ratio was multiplied by a tenderness score of 0 (not tender) or 1 (tender). Tenderness was assessed in the area between the joints. The results of each digit were then added to produce a total score. LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, baseline cDMARD experience, visit, and treatment-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants who had baseline dactylitis, baseline LDI-B score and post baseline LDI-B score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 39 | 23 | 54 | 41
units on a scale | -25.4 (6.53) | -57.1 (7.84) | -57.1 (5.67) | -48.3 (6.31)

20. Secondary Outcome: Change From Baseline in in the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: The BASDAI is a self-administered measure used to answer 6 questions with a 0 to 10 centimeter (cm) VAS pertaining to the 5 major symptoms of axial activity. To give each symptom equal weighting, the mean of the 2 scores relating to morning stiffness was taken. The resulting 0 to 50 score was divided by 5 to give a final 0 to 10 BASDAI Score. BASDAI ranges from 0-10. Higher scores represent greater disease activity. LS mean was calculated using MMRM analysis with treatment, baseline score, geographic region, baseline cDMARD experience, visit, and treatment-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants who had baseline axial involvement defined as baseline BASDAI score >4, baseline BASDAI score and post baseline BASDAI score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 75 | 73 | 85 | 71
units on a scale | -1.25 (0.268) | -2.42 (0.249) | -2.74 (0.234) | -2.91 (0.251)

21. Secondary Outcome: Number of Participants With Treatment Emergent Anti-Ixekizumab Antibodies (TE-ADA) and Neutralizing Antibodies (NAb)
Description: Number of participants with positive treatment emergent anti-ixekizumab antibodies and NAb was summarized by treatment group.
Time Frame: Baseline to Week 24
Population: All randomized participants who received at least 1 dose of ixe and had evaluable anti-ixekizumab antibody measurement at baseline and post baseline or had no evaluable baseline anti-ixekizumab antibody measurements. Immunogenicity data was not collected during the double-blind treatment period for participants in the adalimumab treatment group.
Measure: Number; unit: participants
Arm/Group | Placebo | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 103 | 107 | 100
participants
  Treatment Emergent (TE) | 0 | 6 | 5
  NAb | 0 | 0 | 0

22. Secondary Outcome: Percent Change in American College of Rheumatology-N (ACR-N) Score
Description: The ACR-N score is a continuous measure of clinical, laboratory, and functional outcomes that characterizes the percentage of improvement from baseline in disease activity and the lowest of either a) the percent change in tender joint count (TJC) b) the percent change in swollen joint count (SJC), or c) the median percent change of the remaining 5 ACR core criteria. An ACR-N score of X has improvement of at least X% in both TJC and SJC and a median improvement of at least X% in 5 criteria: patient's assessment of arthritis pain, PatGA, PGA, HAQ-DI and hs-CRP. ACR-N is calculated by allowing for negative results which indicate worsening. LS mean was calculated using Mixed Model Repeated Measurements (MMRM) analysis with treatment, baseline, geographic region, baseline conventional disease modifying anti-rheumatic drugs (cDMARD) experience, visit, and treatment.
Time Frame: Baseline, 24 Weeks
Population: All randomized participants with post-baseline ACR data.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 106 | 101 | 107 | 103
percent change | -4.182 (6.1417) | 28.517 (5.9189) | 33.509 (5.8905) | 30.391 (5.9736)

23. Secondary Outcome: Change From Baseline in Tender Joint Counts (TJC)
Description: TJC is calculated based on tenderness response of 68 joints. TJC possible values range from 0 to 68. A lower TJC indicated less joint tenderness. A higher TJC indicated more joint tenderness. TJC is the number of tender and painful joints determined for each participant by examination of 68 joints. Joints were assessed by pressure and joint manipulation on physical examination. Participants were asked for pain sensations on these manipulations and watched for spontaneous pain reactions. Any positive response on pressure, movement, or both was translated into a single tender-versus-nontender dichotomy. LS mean was calculated using Mixed Model Repeated Measurements (MMRM) analysis with treatment, baseline, geographic region, baseline conventional disease modifying anti-rheumatic drugs (cDMARD) experience, visit, and treatment-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants with baseline and post-baseline TJC data.
Measure: Least Squares Mean (Standard Error); unit: joint counts
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 106 | 100 | 107 | 102
joint counts | -4.7 (1.14) | -10.1 (1.10) | -11.9 (1.08) | -13.6 (1.09)

24. Secondary Outcome: Change From Baseline in Swollen Joint Counts (SJC)
Description: SJC is calculated based on swelling response of 66 joints. SJC possible values range from 0 to 66. A lower SJC indicated less joint swelling. A higher SJC indicated more joint swelling. SJC is the number of swollen joints determined for each participant by examination of 66 joints. Joints were classified as either swollen or not swollen. Swelling was defined as palpable fluctuating synovitis of the joint. LS mean was calculated using Mixed Model Repeated Measurements (MMRM) analysis with treatment, baseline, geographic region, baseline conventional disease modifying anti-rheumatic drugs (cDMARD) experience, visit, and treatment-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants with baseline and post-baseline SJC data.
Measure: Least Squares Mean (Standard Error); unit: joint counts
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 106 | 100 | 107 | 102
joint counts | -3.5 (0.62) | -6.1 (0.59) | -7.0 (0.59) | -8.3 (0.59)

25. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain VAS
Description: The VAS is an instrument used to measure a person's subjective quantitative evaluation of an item such as pain intensity. The VAS contains a continuous line between two end points whereby the respondent places a mark on the line to indicate his or her response. In this study, participants scored their pain intensity in the most affected joint of the gout flare on a 0 100 mm VAS. The scale ranged from 0 (no pain) to 100 (unbearable pain). The scores were measured to the nearest millimeter from the left. LS mean was calculated using Mixed Model Repeated Measurements (MMRM) analysis with treatment, baseline, geographic region, baseline conventional disease modifying anti-rheumatic drugs (cDMARD) experience, visit, and treatment-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants with baseline and post-baseline patient's assessment of pain data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 105 | 99 | 104 | 98
units on a scale | -14.0 (2.68) | -30.0 (2.52) | -29.6 (2.51) | -31.6 (2.54)

26. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Severity (PatGA) VAS
Description: Participants scored their overall assessment of their PsA activity on a 0 to 100 mm horizontal VAS. The scale ranged from 0 (no disease activity) to 100 (extremely active disease activity). The scores were measured to the nearest millimeter from the left. LS mean was calculated using Mixed Model Repeated Measurements (MMRM) analysis with treatment, baseline, geographic region, baseline conventional disease modifying anti-rheumatic drugs (cDMARD) experience, visit, and treatment-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants with baseline and post-baseline patient's global assessment of disease activity data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 105 | 99 | 104 | 98
units on a scale | -14.8 (2.65) | -31.6 (2.49) | -33.8 (2.48) | -35.6 (2.50)

27. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity VAS
Description: The investigator was asked to give an overall assessment of the severity of the participant's current PsA activity using a 0 to 100 mm horizontal VAS. The scale ranged from 0 no disease activity to 100 extremely active disease activity. The scores were measured to the nearest millimeter from the left. Least Square (LS) mean was calculated using Mixed Model Repeated Measurements (MMRM) analysis with treatment, baseline, geographic region, baseline conventional disease modifying anti-rheumatic drugs (cDMARD) experience, visit, and treatment-by-visit interaction.
Time Frame: Baseline, 24 Weeks
Population: All randomized participants with baseline and post-baseline physician's global assessment of disease activity data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 100 | 88 | 96 | 95
units on a scale | -24.2 (2.14) | -34.7 (2.10) | -38.5 (2.06) | -42.0 (1.99)

28. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP)
Description: CRP milligram/liter (mg/L) was measured with a high sensitivity assay at a central laboratory to assess acute phase reactant. LS mean was calculated using Mixed Model Repeated Measurements (MMRM) analysis with treatment, baseline, geographic region, baseline conventional disease modifying anti-rheumatic drugs (cDMARD) experience, visit, and treatment-by-visit interaction.
Time Frame: Baseline, Week 24
Population: All randomized participants with baseline and post-baseline CRP data.
Measure: Least Squares Mean (Standard Error); unit: milligram/liter (mg/L)
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 106 | 101 | 107 | 103
milligram/liter (mg/L) | -3.873 (1.4292) | -7.512 (1.2674) | -8.804 (1.2602) | -8.942 (1.2552)

29. Secondary Outcome: Change From Baseline in Leeds Enthesitis Index (LEI)
Description: as for outcome 8
Time Frame: Baseline, Week 24
Population: All randomized participants who had baseline enthesitis, baseline LEI score and post baseline LEI score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 57 | 56 | 70 | 59
units on a scale | -0.8 (0.26) | -0.9 (0.23) | -1.3 (0.21) | -1.4 (0.24)

30. Secondary Outcome: Percentage of Participants Achieving Psoriasis Area and Severity Index 75%, 90%, 100% (PASI 75, 90, 100)
Description: as for outcome 7
Time Frame: Week 24
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 38 | 61 | 60 | 49
percentage of participants
  PASI 75: number analyzed (Participants) | 7 | 37 | 52 | 45
  PASI 75 | 10.9 | 55.2 | 71.2 | 80.4
  PASI 90: number analyzed (Participants) | 4 | 25 | 41 | 38
  PASI 90 | 6.3 | 37.3 | 56.2 | 67.9
  PASI 100: number analyzed (Participants) | 2 | 16 | 31 | 30
  PASI 100 | 3.1 | 23.9 | 42.5 | 53.6

31. Secondary Outcome: Change From Baseline in Itching Severity Using the Itch NRS
Description: as for outcome 9
Time Frame: Baseline, Week 24
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab Q2W | Ixekizumab Q4W | Ixekizumab Q2W
Number analyzed (Participants) | 67 | 68 | 73 | 59
units on a scale | -0.3 (0.32) | -1.7 (0.29) | -2.9 (0.29) | -2.8 (0.31)

ADVERSE EVENTS:
Description: Adverse events were summarized based on all randomized participants who received at least one dose of study drug.
Groups:
- Placebo (PBO) Double-Blind Period: Participants received placebo for ixekizumab (ixe) as 2 subcutaneous (SC) injections and placebo for adalimumab as one SC injection for a total of 3 injections at Week 0. Placebo for ixekizumab and placebo for adalimumab were given as single SC injections every 2 weeks (Q2W) from Week 2 to Week 24.
- Adalimumab (ADA) Double-Blind Period; IR IXE Q4W: Participants received 40 mg of adalimumab as one SC injection and placebo for ixekizumab as 2 SC injections for a total of 3 injections at Week 0. Participants received one SC injection of 40 mg of adalimumab and one SC injection of placebo for ixekizumab Q2W from Week 2 to Week 24
- Ixe Q2W Double-Blind Period; IR IXE Q2W: Participants received a starting dose of 160 mg of ixekizumab given as 2 SC injections of 80 mg and placebo for adalimumab as one SC injection for a total of 3 injections at Week 0. Participants received one SC injection of 80 mg of ixekizumab or placebo for ixekizumab Q2W from Week 2 to Week 24. Participants received one SC injection of placebo for adalimumab Q2W from Week 2 to Week 24.
- Ixe Q4W Double-Blind Period: Participants received a starting dose of 160 mg of ixekizumab given as 2 SC injections of 80 mg and placebo for adalimumab as one SC injection for a total of 3 injections at Week 0. Participants received one SC injection of 80 mg of ixekizumab Q2W or Placebo for ixekizumab (ixe) Q2W from Week 2 to Week 24. Participants received one SC injection of placebo for adalimumab Q2W from Week 2 to Week 24.
- IR PBO Washout: Participants received placebo for ixekizumab as 2 SC injections and placebo for adalimumab as one SC injection for a total of 3 injections at Week 0. Placebo for ixekizumab and placebo for adalimumab were given as single SC injections Q2W from Week 2 to Week 24.
- PBO Washout: Participants received a starting dose of 160 mg of ixekizumab given as 2 SC injections of 80 mg and placebo for adalimumab as one SC injection for a total of 3 injections at Week 0. Participants received one SC injection of 80 mg of ixekizumab Q2W from Week 2 to Week 24. Participants received one SC injection of placebo for adalimumab Q2W from Week 2 to Week 24.
- IXE Q4W: Ixekizumab every 4 weeks (IxeQ4W) and IR IxeQ4W participants received one SC injection of 80 mg of alternating ixekizumab or placebo for ixekizumab Q2W from Week 24 to Week 156.
  Placebo and IR placebo (PBO) Washout participants re-randomized to Ixekizumab 80 mg Q4W received a starting dose of 160 mg of ixekizumab given as 2 SC injections of 80 mg and placebo for adalimumab as one SC injection for a total of 3 injections at Week 24. Participants received one SC injection of 80 mg of alternating placebo for ixekizumab or ixekizumab Q2W from Week 26 to Week 156.
  PBO Washout participants re-randomized to ixekizumab 80 mg Q4W received one SC injection of 80 mg of alternating ixekizumab or placebo for ixekizumab Q2W from Week 32 to Week 156.
- IXE Q2W: Ixekizumab Q2W (IxeQ2W) and IR IxeQ2W participants received one SC injection of 80 mg of ixekizumab Q2W from Week 24 to Week 156.
  Placebo and IR PBO Washout participants re-randomized to Ixekizumab 80 mg Q2W received a starting dose of 160 mg of ixekizumab given as 2 SC injections of 80 mg and placebo for adalimumab as one SC injection for a total of 3 injections at Week 24. Participants received one SC injection of 80 mg of ixekizumab Q2W from Week 26 to Week 156.
  PBO Washout participants re-randomized to ixekizumab 80 mg Q2W received one SC injection of 80 mg of ixekizumab Q2W from Week 32 to Week 156.
- PBO Post-Treatment Follow-Up Period: Participants discontinued the study early and entered the post-treatment follow-up period. Participants received placebo immediately prior to entering the post-treatment follow-up period.
- IXE Q4W Post-Treatment Follow-up Period: Participants either completed the study or discontinued the study early and entered the post-treatment follow-up period. Participants received ixekizumab 80 mg Q4W immediately prior to entering the post-treatment follow-up period.
- IXE Q2W Post-Treatment Follow-up Period: Participants either completed the study or discontinued the study early and entered the post-treatment follow-up period. Participants received ixekizumab 80 mg Q2W immediately prior to entering the post-treatment follow-up period.
Arm/Group | Placebo (PBO) Double-Blind Period | Adalimumab (ADA) Double-Blind Period | Ixe Q2W Double-Blind Period | Ixe Q4W Double-Blind Period | IR IXE Q4W | IR IXE Q2W | IR PBO Washout | PBO Washout | IXE Q4W | IXE Q2W | PBO Post-Treatment Follow-Up Period | Adalimumab Post-Treatment Follow-up Period | IXE Q4W Post-Treatment Follow-up Period | IXE Q2W Post-Treatment Follow-up Period
Serious Adverse Events (participants affected / at risk) | 2/106 | 5/101 | 6/107 | 3/102 | 0/24 | 0/24 | 0/9 | 1/88 | 28/187 | 19/183 | 0/20 | 0/1 | 2/165 | 2/171
Other Adverse Events (participants affected / at risk) | 16/106 | 18/101 | 33/107 | 31/102 | 0/24 | 0/24 | 0/9 | 7/88 | 62/187 | 66/183 | 0/20 | 0/1 | 0/165 | 0/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (PBO) Double-Blind Period (N=106) | Adalimumab (ADA) Double-Blind Period (N=101) | Ixe Q2W Double-Blind Period (N=107) | Ixe Q4W Double-Blind Period (N=102) | IR IXE Q4W (N=24) | IR IXE Q2W (N=24) | IR PBO Washout (N=9) | PBO Washout (N=88) | IXE Q4W (N=187) | IXE Q2W (N=183) | PBO Post-Treatment Follow-Up Period (N=20) | Adalimumab Post-Treatment Follow-up Period (N=1) | IXE Q4W Post-Treatment Follow-up Period (N=165) | IXE Q2W Post-Treatment Follow-up Period (N=171)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Latent tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/48 (0) | 0/51 (0) | 0/45 (0) | 0/47 (0) | 0/8 (0) | 0/8 (0) | 0/1 (0) | 0/50 (0) | 0/78 (0) | 0/92 (0) | 0/10 (0) | 0 (0) | 0/71 (0) | 1/87 (1)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Guillain-barre syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acquired phimosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bartholin's cyst (Reproductive system and breast disorders) | 1/58 (1) | 0/50 (0) | 0/62 (0) | 0/55 (0) | 0/16 (0) | 0/16 (0) | 0/8 (0) | 0/38 (0) | 0/109 (0) | 0/91 (0) | 0/10 (0) | 0 (0) | 0/94 (0) | 0/84 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0/58 (0) | 1/50 (1) | 0/62 (0) | 0/55 (0) | 0/16 (0) | 0/16 (0) | 0/8 (0) | 0/38 (0) | 0/109 (0) | 0/91 (0) | 0/10 (0) | 0 (0) | 0/94 (0) | 0/84 (0)
Uterine polyp (Reproductive system and breast disorders) | 0/58 (0) | 0/50 (0) | 1/62 (1) | 0/55 (0) | 0/16 (0) | 0/16 (0) | 0/8 (0) | 0/38 (0) | 0/109 (0) | 0/91 (0) | 0/10 (0) | 0 (0) | 0/94 (0) | 0/84 (0)
Vulval disorder (Reproductive system and breast disorders) | 0/58 (0) | 0/50 (0) | 0/62 (0) | 0/55 (0) | 0/16 (0) | 0/16 (0) | 0/8 (0) | 0/38 (0) | 1/109 (1) | 0/91 (0) | 0/10 (0) | 0 (0) | 0/94 (0) | 0/84 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (PBO) Double-Blind Period (N=106) | Adalimumab (ADA) Double-Blind Period (N=101) | Ixe Q2W Double-Blind Period (N=107) | Ixe Q4W Double-Blind Period (N=102) | IR IXE Q4W (N=24) | IR IXE Q2W (N=24) | IR PBO Washout (N=9) | PBO Washout (N=88) | IXE Q4W (N=187) | IXE Q2W (N=183) | PBO Post-Treatment Follow-Up Period (N=20) | Adalimumab Post-Treatment Follow-up Period (N=1) | IXE Q4W Post-Treatment Follow-up Period (N=165) | IXE Q2W Post-Treatment Follow-up Period (N=171)
Injection site erythema (General disorders) | 0 (0) | 2 (5) | 7 (11) | 13 (42) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 5 (51) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 3 (5) | 13 (31) | 16 (63) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 12 (63) | 13 (180) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 4 (5) | 3 (3) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (13) | 10 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (7) | 12 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 5 (5) | 5 (5) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 21 (27) | 18 (23) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 5 (6) | 6 (7) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 21 (32) | 21 (23) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (11) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days